CLINICAL TRIAL: NCT00063011
Title: Calcium and Exercise Effect on Pubertal Bone Gain
Brief Title: Bone Development in Adolescent Girls: Effects of Calcium and Exercise
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01HD036601 (NIH)
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Osteoporosis
Keywords: Weight-bearing exercise; Calcium-rich diet; Adolescents; Females; Bone mass; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Resistance Training

INTERVENTIONS:
Behavioral: Calcium rich diet
Behavioral: Weight bearing exercise

SUMMARY:
Osteoporosis is a major public health problem. Prevention of osteoporosis depends in part on good bone development in childhood and adolescence. This study will evaluate a weight-bearing exercise program and high-calcium diet on bone development in adolescent girls.

DETAILED DESCRIPTION:
There are currently few safe and effective methods for restoring lost bone to the osteoporotic skeleton. Therefore, prevention of osteoporosis is crucial. If skeletal development can be maximized during growth, young people will begin adulthood with optimal bone mass and will be less likely to develop osteoporosis in later years. This study will determine the effects of weight-bearing physical activity and a high-calcium diet on bone mass in adolescent girls.

Participants in this study will be randomized to one of three study arms. Girls in Arm 1 will consume their usual diets and will participate in a weight-bearing exercise program that meets 3 times per week. Girls in Arm 2 will also participate in a weight-bearing exercise program that meets 3 times per week and will be given high calcium foods to supply 1500 mg of calcium per day. Girls in Arm 3 will consume their usual diet and maintain their customary activity level. Study visits occur every 6 months; participants will be followed for 4 ½ years. Assessments will include a medical and social history and measurements of spine, hip, radius, and total body bone mineral content (BMC); calcaneal speed of sound (SOS); height; weight; and Tanner stage.

ELIGIBILITY:
Inclusion Criteria

* Tanner Stage of Development: Stage 1

Exclusion Criteria

* History of lactose intolerance, milk allergy, corticosteroid or anticonvulsant therapy, familial hypercholesterolemia, mental or physical handicaps, cancer, rheumatoid arthritis, asthma, or any other significant health problem
* Body mass index (BMI) >= 85th percentile for age and gender
* Regularly have more than two practice sessions per week of dance, gymnastics, or organized team sports

Ages: 9 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 107
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Joan M. Lappe, Ph.D., Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States